CLINICAL TRIAL: NCT06619821
Title: Effects of Parent-Adolescent Joint Interventions for Adolescents With Adverse Childhood Experiences: A Multi-Center Cluster Randomized Controlled Trial
Brief Title: Effects of Parent-Adolescent Joint Interventions for Adolescents With Adverse Childhood Experiences
Acronym: EASY-PEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Joint Tx for Adolscents ACEs
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Stress, Emotional; Stress-related Mental Disorders; Adverse Childhood Experiences
Keywords: adolescents; randomized controlled trial; PTSD; ACE; depression; anxiety
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psychoeducation group （PsyE） (Active Comparator): Psychoeducation consists of parent and adolescent psychoeducation. The content includes an introduction to stress, emotional distress and mental disorders.
  Interventions: Behavioral: Psychoeducation
- Psychoeducation + Emotional Skills (PsyE+EmoS) (Experimental): Psychoeducation includes sessions for both parents and adolescents, offering the same content as the control group, which introduces stress, emotional distress, and mental disorders.
  In addition, the emotional skills enhancement sessions provide online materials focused on emotional awareness and emotion regulation strategies, along with tasks related to the content. Participants will also be required to complete a weekly writing assignment, upload their written contents, and assess their level of subjective discomfort following each writing exercise.
  Interventions: Behavioral: Emotiaonl skill enhancement; Behavioral: PCE promotion; Behavioral: Psychoeducation
- Psychoeducation + emotional skills + PCE (PsyE+EmoS+PoCE) (Experimental): In comparison to the PsyE+EmoS group, this group additionally requires parents to complete a weekly parent-child communication task aimed at fostering positive childhood experiences. Parents are also expected to document and upload the details of these tasks each week.
  Interventions: Behavioral: Emotiaonl skill enhancement; Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Emotiaonl skill enhancement — This intervention combines online material with practical, emotion-focused activities. Participants will receive training on emotional awareness and emotion regulation strategies, along with completing weekly writing assignments. These assignments focus on recent negative events and the emotions associated with them, encouraging emotional expression and processing.
  Arms: Psychoeducation + Emotional Skills (PsyE+EmoS); Psychoeducation + emotional skills + PCE (PsyE+EmoS+PoCE)
Behavioral: PCE promotion — The intervention requires parents to complete a weekly parent-child interaction task designed to foster positive childhood experiences. Parents will engage in structured activities with their children and document the interactions. Each week, they are expected to upload a report.
  Arms: Psychoeducation + Emotional Skills (PsyE+EmoS)
Behavioral: Psychoeducation — Psychoeducation includes sessions for both parents and adolescents, covering key topics such as stress, emotional distress, and mental disorders. The content provides foundational knowledge to help participants understand and manage these challenges.

SUMMARY:
The study aims to examine the effectiveness of joint parent-adolescent intervention in improving the mental health outcomes of participants, specifically by reducing symptoms of depression, anxiety, and PTSD, as measured by the Patient Health Questionnaire (PHQ-9), the Generalized Anxiety Disorder-7 scale (GAD-7), and the Child PTSD Symptom Scale for DSM-5 (CPSS-5). Adolescents will be recruited from middle schools and randomly assigned to one of three groups: (a) psychoeducation, (b) psychoeducation + emotional skills enhancement, or (c) psychoeducation + emotional skills enhancement + positive childhood experience promotion. The school-based intervention will consist of 4-8 sessions, with assessments conducted at baseline, post-treatment, and a 3-month follow-up. Investigators will conduct multilevel models (MLMs) and structural equation models (SEMs) to investigate the impact of Adverse Childhood Experiences (ACEs), Positive Childhood Experiences (PCEs), alexithymia, and emotion regulation abilities on mental health outcomes in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Middle school students studying in school and their parents
* Capable of hearing, speaking, reading, and writing

Exclusion Criteria:

* High suicidal risks
* Severe mental disorders

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Alexithymia | baseline, post treatment(1 month), 3 month after post treatment
  A 36-item Peking alexithymia scale measures thoughts and behaviors that prevent people from feeling or recognizing negative emotions on a 5-point Likert scale (1 to 5, and total scores vary from 36 to 180). A higher score represents more severe alexithymia.
PTSD for adolescents | baseline, post treatment(1 month), 3 month after post treatment
  The Child PTSD Symptom Scale for DSM-5 (CPSS-5) for adolescents and children (scores from 0 to 4, and total scores vary from 0 to 80). A higher score represents worse PTSD symptoms.
Emotion awareness | baseline, post treatment(1 month), 3 month after post treatment
  A 30-item Emotion awareness questionnaire measures emotion awareness on a 3-point Likert scale (1 to 3, and total scores vary from 30 to 90). A higher score represents better emotion awareness.
Emotion regulation | baseline, post treatment(1 month), 3 month after post treatment
  An 18-item cognitive emotion regulation questionnaire measures the ability of emotion regulation on a 5-point Likert scale (1 to 5, and total scores vary from 18 to 90). A higher score represents better emotion regulation.
Depression | baseline, post treatment(1 month), 3 month after post treatment
  The 9-item patient health questionnaire (PHQ-9) for adults (score from 0 to 3, and total score varies from 0 to 27). A higher score represents worse depression symptoms.
Generalized anxiety disorder | baseline, post treatment(1 month), 3 month after post treatment
  The Generalized Anxiety Disorder-7 scale (GAD-7) for adults, adolescents, and children (scored from 0 to 3, and total score from 0 to 21). A higher score represents worse anxiety symptoms.

SECONDARY OUTCOMES:
Irritability | baseline, post treatment(1 month), 3 month after post treatment
  A 17-item irritability measurement scale, the Peking irritability scale, measures impulsive emotions, thoughts, and behaviors on a 5-point Likert scale (score from 1 to 5, and total score varies from 17 to 85). A higher score represents higher irritability.
Resilience | baseline, post treatment(1 month), 3 month after post treatment
  A 10-item resilience measurement scale, the Connor-Davidson resilience scale, measures resilience on a 5-point Likert scale (score from 0 to 4, and total score varies from 0 to 40). A higher score represents better resilience .
Seeking for help | baseline, post treatment(1 month), 3 month after post treatment
  A 10-item help-seeking scale measures on a 7-point Likert scale (score from 1 to 7, and total score varies from 10 to 70), with higher scores indicating greater willingness to seek help from others.
Insomnia Severity | baseline, post treatment(1 month), 3 month after post treatment
  The severity of insomnia symptoms will be assessed using the Insomnia Severity Index (ISI). This 7-item self-report measurement evaluates the severity of insomnia symptoms, the level of satisfaction with sleep, interference with daily functioning, noticeability of impairment attributed to sleep problems, and the level of distress caused by sleep disturbance (score from 0 to 4, and total score vary from 0 to 32). Each item is rated on a 5-point scale, providing a comprehensive measure of insomnia severity.

OTHER OUTCOMES:
Suicide | baseline, post treatment(1 month), 3 month after post treatment
  The suicidal behaviors questionnaire-revised (SBQ-R) for adolescents and children (total scores vary from 3 to 18). A higher score represents a higher suicide risk.
Self-esteem | baseline, post treatment(1 month), 3 month after post treatment
  A 10-item self-esteemmeasurement scale, Rosenberg self-esteem scale, measures self-esteem on a 4-point Likert scale (score from 0 to 3, and total score varies from 0 to 30), with higher scores indicating greater self-esteem.
Social support | baseline, post treatment(1 month), 3 month after post treatment
  The 12-item Multidimensional Scale of Perceived Social Support (score from 1 to 7, and total score varies from 12 to 84). A higher score represents better social support.
Subjective Happiness Scale | baseline, post treatment(1 month), 3 month after post treatment
  A 4-item subjective happiness scale measures happiness (score from 1 to 7, and total score vary from 4 to 28). A higher score represents a happier state.
Subjective Units of Distress Scale | each week during intervention (up to 4 months)
  A single item inquires about subjective distress on a 100-point scale. A higher score represents more subjective distress.
Positive Childhood Experiences | baseline, post treatment(1 month), 3 month after post treatment
  A questionnaire measuring positive childhood experiences with 13 items(total scores vary from 0 to 64). A higher score represents a more positive childhood experiences.
Game Addiction Scale | baseline, post treatment(1 month), 3 month after post treatment
  A 7-item game addiction scale, measures game addiction on a 5-point Likert scale (score from 1 to 5, and total score varies from 7 to 35), with higher scores indicating worse game addiction.
Behavior performances | baseline, post treatment(1 month), 3 month after post treatment
  A 22-item behavior performance questionnaire measures various behavior performances such as study time, phone use, school performance, drinking alcohol, smoking, stealing, fighting, and lying.
Adverse events | baseline, post treatment(1 month)
  A 33-item adverse events questionnaire asks about adverse events before 18, including self-harm, experiencing emotional abuse, experiencing physical abuse, feeling severe distress, mental illness events (e.g., panic attack), and physical injury, etc. The score of each item ranges from 0 to 1(0=no, 1=yes), 0 to 4, or 0 to 5 (a higher score indicates a more severe adverse event)
Meaning in life | baseline, post treatment(1 month), 3 month after post treatment
  A 6-item meaning in life scale measures life meaning (score from 1 to 5, and total score vary from 6 to 30). A higher score represents more life meaning perception.
Non-suicidal self-injury | baseline, post treatment(1 month), 3 month after post treatment
  The non-suicidal self-injury assessment tool (NSSI-AT-Severity) for adolescents and children (total scores vary from 5 to 16). A higher score represents a worse self-injury situation.
Self-esteem stability | baseline, post treatment(1 month), 3 month after post treatment
  A 5-item Labile Self-Esteem Scale measures self-esteem stability on a 5-point Likert scale (score from 1 to 5, and total score varies from 5 to 25), with lower scores indicating better self-esteem stability.
Somatic problems | baseline, post treatment(1 month), 3 month after post treatment
  A somatic problems scale modified from PHQ-15, measuring various physical discomforts and pain on a 3-point Likert scale (score from 0 to 2). A higher score represents worse somatic problems.
Problematic Internet use | baseline, post treatment(1 month), 3 month after post treatment
  A 10-item problematic Internet use scale measures problematic Internet use on a 7-point Likert scale (score from 1 to 7, and total score varies from 7 to 49), with higher scores indicating greater problematic Internet use.
Adverse Childhood Experiences | baseline, post treatment(1 month), 3 month after post treatment
  An adverse childhood experiences questionnaire measuring the adverse childhood experiences with 26 items. A higher number of adverse childhood experiences represents worse childhood experiences.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Biancun middle school, Baoding, Hebei
  - Diannan middle school, Baoding, Hebei

IPD SHARING:
Plan to Share IPD: Undecided